CLINICAL TRIAL: NCT03237052
Title: A Randomized Controlled Multi-center Clinical Study Focusing on Validating and Optimizing Model of Antipsychotics Selection in China
Brief Title: Validating and Optimizing Model of Antipsychotics Selection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VOMAS-C
Record Dates: First submitted 2017-07-29; First posted 2017-08-02 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Models, Biological; Nonlinear Dynamics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- model (Experimental): model aided decision
  Interventions: Other: model
- non-model (Active Comparator): real-world psychiatrist decision
  Interventions: Other: non-model

INTERVENTIONS:
Other: model — a model that has been established in advance.
  Other Names: model aided decision
  Arms: model
Other: non-model — real-world psychiatrist decision
  Other Names: non-model decision
  Arms: non-model

SUMMARY:
This multi-centre study will evaluate the clinical efficacy of 3 atypical antipsychotics treatment in Chinese Patients with Schizophrenia by comparing model-decision with real-world psychiatrist-decision. The three atypical antipsychotics are olanzapine (5-20 milligram per day), risperidone (2-6 milligram per day) and aripiprazole (5-30 milligram per day). The main purpose of this study is to explore the potential difference between modal-aided-decision with clinician-decision in order to validate and optimize the selection model that has been established in advance.

The efficacy evaluations include symptoms, social function, recurrence rate and hospitalization. Visits occurs at 0, 4, 8, 13, 26, 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* An in-patient or out-patient (male or female) and aged ≥18 years
* A diagnosis of schizophrenia, DSM-5 (Diagnostic and Statistical Manual Diploma in Social Medicine-5)
* Subjects must have the ability to effectively communicate with investigator, complete study related documents, comprehend the key components of the consent form and must provide written informed consent to participate in the study prior to any study specific assessments or procedures.
* Patients are taking or will take atypical antipsychotics which include olanzapine, risperidone, aripiprazole.
* Baseline PANSS Total Score ≥70

Exclusion Criteria:

* Participation in other clinical studies.
* Known intolerance or lack of efficacy to olanzapine, risperidone or aripiprazole.
* Use of clozapine within 28 days prior to randomization.
* Other conditions which, in the investigator's judgment, render patients unsuitable for the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of PSP from Baseline | 52 weeks
  PSP assessment at 52 weeks

SECONDARY OUTCOMES:
Change of PANSS from Baseline | 52 weeks
  PANSS assessment at 52 weeks
Change of CDSS from Baseline | 52 weeks
  CDSS assessment at 52 weeks
Change of CGI from Baseline | 52 weeks
  CGI assessment at 52 weeks
Change of liver function from Baseline | 52 weeks
  Liver function assessment at 52 weeks
Change of PRL from Baseline | 52 weeks
  PRL assessment at 52 weeks
Number of Participants with EPS | 52 weeks
  EPS assessment at 52 weeks
Number of Participants with abnormal ECG | 52 weeks
  ECG assessment at 52 weeks
Number of Participants with abnormal sexual function | 52 weeks
  sexual function assessment at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng SHEN, MD PhD, Principal Investigator — GCP Office
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No